CLINICAL TRIAL: NCT04987970
Title: An Open Label, Randomized, Single Dose, 2-sequence, 4-period, Cross-over Clinical Trial to Evaluate the Pharmacokinetics and Tolerability of CKD-386(2) With Co-administration of D013, D326, and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of CKD-386(2) 80/20/10mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A83_07BE2117
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-12

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: D013, D326, D337- A single oral dose of 3 tablets under fasting condition Period 2: CKD-386(2)- A single oral dose of 1 tablet under fasting condition Period 3: D013, D326, D337- A single oral dose of 3 tablets under fasting condition Period 4: CKD-386(2)- A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-386(2); Drug: D013, D326, D337
- Sequence 2 (Experimental): Period 1: CKD-386(2)- A single oral dose of 1 tablet under fasting condition Period 2: D013, D326, D337- A single oral dose of 3 tablets under fasting condition Period 3: CKD-386(2)- A single oral dose of 1 tablet under fasting condition Period 4: D013, D326, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-386(2); Drug: D013, D326, D337

INTERVENTIONS:
Drug: CKD-386(2) — QD, PO
Drug: D013, D326, D337 — QD, PO

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and Tolerability of CKD-386(2)

DETAILED DESCRIPTION:
An open label, randomized, single dose, 2-sequence, 4-period, cross-over clinical trial to evaluate the pharmacokinetics and tolerability of CKD-386(2) with co-administration of D013, D326, and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who meet the blood pressure criteria during screening tests:

   * Systolic Blood Pressure: 90 to 139 mmHg
   * Diastolic Blood Pressure: 60 to 89 mmHg
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory(hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial.
7. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month before the first administration of investigational products.
3. Those who donated whole blood or apheresis within 8 weeks or 4 weeks respectfully, or received blood transfusion within a 4 weeks.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption than below criteria

   * Alcohol: Man_21 glasses/week, Woman_14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL)
   * Heavy Smoking: 20 cigarettes/day
6. Patients with the following diseases

   * Patients with hypersensitivity to the main constituents or components of the investigational drug
   * Severe hepatic impairment, biliary atresia or cholestasis
   * Patients with hereditary angioedema or with a history of angioedema in the treatment of ACE inhibitors or angiotensin II receptor antagonists
   * Diabetes mellitus
   * Patients with moderate to severe renal impairment [glomerular filtration rate (eGFR) <60 mL / min / 1.73m^2]
   * Renal vascular hypertension patients
   * Patients with active liver disease, including unexplained persistent serum transaminase elevations or elevated serum transaminase elevations greater than three times the normal upper limit
   * Patients with myopathy or have a history of family or genetic history of myopathy
   * Hypothyroidism
   * If you have a history of muscle toxicity for other HMG-CoA converting enzymes or fibrate class drugs
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Area under the concentration-time curve from time zero to time
Cmax of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Area under the concentration-time curve from zero up to ∞
Tmax of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Time to maximum plasma concentration
AUCt/AUCinf of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  AUCt/AUCinf
T1/2 of CKD-386(2) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D., PhD., Principal Investigator — Seoul, Gwanak-gu, South Korea, 08779
Locations (1):
- H plus Yangji hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No